CLINICAL TRIAL: NCT01047488
Title: Randomised, Double-blind, Placebo-controlled Trial of the Effect of the Combination of Imipramine and Pregabalin for the Treatment of Painful Polyneuropathy
Brief Title: Imipramine and Pregabalin Combination in Painful Polyneuropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Pfizer (Industry); Nycomed (Industry)
Responsible Party: Søren Hein Sindrup, Department of Neurology, Odense University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tcapgbcomb1; 2009-013642-80 (EudraCT Number)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Polyneuropathy
Keywords: polyneuropathy; neuropathic pain; treatment
MeSH Terms: conditions — Polyneuropathies; Neuralgia | interventions — Imipramine; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Imipramine (Active Comparator): Imipramine tablets and placebo capsules to pregabalin
  Interventions: Drug: Imipramine
- Pregabalin (Active Comparator): Pregabalin capsules and placebo tablets to imipramine
  Interventions: Drug: Pregabalin
- Imipramine plus pregabalin (Experimental): Imipramine tablets and pregabalin capsules
  Interventions: Drug: Imipramine, pregabalin
- Placebo (Placebo Comparator): Placebo tablets to imipramine and placebo capsules to pregabalin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imipramine — Tablet 25 mg, 3 tablets evening (extensive metabolizers) or 1 tablet evening (poor metabolizers), daily, 5 weeks
  Other Names: Imipramin DAK
  Arms: Imipramine
Drug: Pregabalin — Capsule 75 mg, 2 capsules twice daily, daily, 5 weeks
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Imipramine, pregabalin — Imipramine: tablet 25 mg, 3 tablets evening (extensive metabolizers) or 1 tablet evening (poor metabolizers), daily, 5 weeks Pregabalin: capsule 75 mg, 2 capsules twice daily, daily, 5 weeks
  Other Names: Imipramin DAK; Lyrica
  Arms: Imipramine plus pregabalin
Drug: Placebo — Placebo tablets to imipramine 25 mg, 3 or 1 tablet evening, daily, 5 weeks Placebo capsules to pregabalin 75 mg, 2 capsules daily, daily, 5 weeks
  Arms: Placebo

SUMMARY:
Polyneuropathy of different etiologies is often associated with pain and the standard treatment for this type of pain is gabapentinoids or antidepressants. The hypothesis of this study is that the combination of the gabapentinoid pregabalin and the antidepressant imipramine will provide better pain relief than the single compounds alone.

This is a randomized, placebo-controlled, double-blind, 4-way, cross-over trial of pregabalin 300 mg/day, imipramine 75 mg/day and their combination versus placebo. The study will include 60 patients and the treatment outcome will be pain intensity as measured by numeric rating scales.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 - 85 years.
* Characteristic symptoms of polyneuropathy for at least 6 months.
* Polyneuropathy diagnosis confirmed by typical clinical signs (distal sensory disturbance/lack of distal deep tendon reflexes) and/or electrophysiological tests and/or abnormal quantitative sensory tests.
* Total pain intensity rating of at least 4 on a 0-10 points numeric rating scale.
* Pain present at least 4 days a week.
* For diabetics: diabetes diagnosis for at least 6 months and stable metabolic control for at least 3 months.
* For other secondary polyneuropathies: stable for at least 6 months.
* For fertile females: adequate anticonceptive treatment.
* Written informed consent.

Exclusion Criteria:

* Other cause of pain.
* Contraindications against imipramine.
* Allergic reactions towards imipramine or pregabalin.
* Known adverse reactions during imipramine or pregabalin treatment.
* Pregnancy.
* Severe systemic disease.
* Ongoing treatment with antidepressants, antipsychotics, anticonvulsants, opioids, propranolol, kinidine, monoamine oxidase inhibitor.
* Inability to follow study protocol.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Total pain intensity as measured by numeric rating scale 0-10 points. | Median of ratings from last week of each treatment period

SECONDARY OUTCOMES:
Verbal pain relief scale with 6 classes | End of each treatment period
Specific pain symptom rated by numeric rating scales 0-10 points | Median of ratings from last week of each treatment period
Rating of evoked pains symptoms (pressure, brush, repetitive pin-prick, cold) as measured by numeric rating scales 0-10 points | End of each treatment period
Sleep disturbance as measured by numeric rating scale 0-10 points | Median of ratings from last week of each treatment period
Consumption of escape medication (number of tablets of paracetamol) | Total consumption during last week of each treatment period
Health related quality of life (SF-36) | End of each treatment period
Major Depression Inventory (MDI) | End of each treament period

CONTACTS AND LOCATIONS:
Overall Officials: Søren H. Sindrup, MD, Study Chair — Department of Neurology, Odense University Hospital; Jakob V. Holbech, MD, Principal Investigator — Department of Neurology, Odense University Hospital
Locations (3):
- Denmark (3):
  - Department of Neurology, Aalborg Hospital, Aalborg
  - Department of Neurology, Aarhus University Hospital, Aarhus
  - Department of Neurology, Odense University Hospital, Odense